CLINICAL TRIAL: NCT00695058
Title: Transcutaneous Mechanical Nerve Stimulation (TMNS) by Vibration in the Treatment of Incontinence
Acronym: TMNS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure to include
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Mikkel Fode/medical student, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-B-2007-047
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Urinary Incontinence
Keywords: Stress incontinence; urge incontinence; overactive bladder syndrome; vibration; nerve stimulation
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): Women with stress incontinence treated with active TMNS (vibration)
  Interventions: Device: Transcutaneous mechanical nerve stimulation by A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Danmark)
- 2 (Placebo Comparator): Women with stress incontinence treated with placebo TMNS (vibration)with an amplitude of 0
  Interventions: Device: Transcutaneous mechanical nerve stimulation by A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Danmark)
- 3 (Experimental): Women with overactive bladder syndrome treated with active TMNS (vibration)
  Interventions: Device: Transcutaneous mechanical nerve stimulation by A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Danmark)
- 4 (Placebo Comparator): Women with overactive bladder syndrome treated with placebo TMNS (vibration)with an amplitude of 0
  Interventions: Device: Transcutaneous mechanical nerve stimulation by A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Danmark)
- 5 (Experimental): males who are still incontinent at a minimum of one year after a radical prostatectomy treated with active TMNS (vibration)
  Interventions: Device: Transcutaneous mechanical nerve stimulation by A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Danmark)
- 6 (Placebo Comparator): males who are still incontinent at a minimum of one year after a radical prostatectomy treated with placebo TMNS (vibration)with an amplitude of 0
  Interventions: Device: Transcutaneous mechanical nerve stimulation by A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Danmark)

INTERVENTIONS:
Device: Transcutaneous mechanical nerve stimulation by A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Danmark) — A medical vibrator (FERTI CARE personel, Multicept A/S, Albertslund, Denmark) will be used. The stimulation works through a vibrating disc of hard plastic with a diameter of 3.5 cm. The stimulation point will be the perineum in women and the perineum or the frenulum in men.
  In the women the stimulation will be performed with a vibration amplitude of 2 mm and a frequency of 100 Hz. In the men the vibration parameter/location will be determined by the results of the new pressure profile studies (aim 3).
  A daily stimulation sequence consisting of 10 seconds of stimulation followed by a 10 second pause repeated 10 times will be used through 6 weeks in both the women with stress incontinence and overactive bladder syndrome.
  In the 3 groups of patients the subjects will be randomized to either active treatment or placebo treatment. The placebo treatment will be done with a vibration device with an amplitude of 0 mm. Subjects will be randomized by a draw.

SUMMARY:
During transcutaneous mechanical nerve stimulation in spinal cord injured men an increase in pressure was observed in the external urethral sphincter along with an increase in bladder capacity. In a subsequent study it was demonstrated that TMNS in women could induce pressure increment of the external urethral sphincter. A pilot study have since shown that after 6 weeks of stimulation 24 out of 33 women suffering from urinary stress incontinence were able to contract their pelvic floor muscles and had become free of symptoms. Another pilot study has shown promising effect on the overactive bladder syndrome.

The present study aims to treat urinary incontinence and includes 3 groups of patients with 40 patients in each group: Women suffering from urinary stress incontinence, women suffering from urge incontinence and men suffering from urinary incontinence after a prostatectomy. A medical vibrator is used and in each group the subjects will be randomized to active treatment or placebo treatment.

In women the stimulation will be performed at the perineum every day for 6 weeks with an amplitude of 2 mm and a frequency of 100 Hz. In men the vibration parameter/location will be determined by the results of a pressure profile study also included. Results will be evaluated on the basis of questionnaires, micturition diaries and diaper tests.

If we are able to demonstrate a significant reduction in the incontinence symptoms in the subjects we asses that vibration can be a way of reestablishing a normal function of the pelvic floor muscles and bladder function in incontinent patients.

ELIGIBILITY:
Inclusion Criteria:

* Women suffering from stress incontinence
* Women suffering from overactive bladder syndrome
* Men who are still incontinent at a minimum of one year after a radical prostatectomy

Exclusion Criteria:

* Pregnant and nursing women will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Diaper test - weight (grams); Micturition diary - The number of involuntary incontinence and normal micturition episodes; Amplitude of vibration (mm) and pressure (cm H2O) in the external sphincter of the urethra | Before treatment, after treatment and at follow up

SECONDARY OUTCOMES:
Validated symptom score (ICI-Q) including: changes in incontinence and micturition patterns; patients' subjective assessment of their symptoms | before treatment, after treatment and at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Sonksen, MD, Ph.D, Study Director — Copenhagen University Hospital at Herlev
Locations (3):
- Department of Urology, University of Michigan, Ann Arbor, Michigan, United States
- Denmark (2):
  - Department of Urology, Herlev University Hospital, Herlev
  - The Regional Hospital of Viborg, Viborg